CLINICAL TRIAL: NCT04786379
Title: Open vs Arthroscopic Treatment of Septic Arthritis in the Adult Native Knee: A Prospective Trial
Brief Title: Surgical Management of Knee Septic Arthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of adequate patient sample size in a reasonable time period and lack of research support staff
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Matthew Wells, Principal Investigator, Texas Tech University Health Sciences Center, El Paso
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #E21085
Record Dates: First submitted 2021-02-24; First posted 2021-03-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Septic Arthritis
Keywords: orthopedic; septic arthritis; synovectomy
MeSH Terms: conditions — Arthritis, Infectious | interventions — Debridement; Therapeutic Irrigation

STUDY DESIGN:
Intervention Model Description: Patients who are diagnosed with septic arthritis of the native knee will be randomized to either arthroscopic or open treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with confirmed septic arthritis of the native knee (Experimental)
  Interventions: Procedure: Arthroscopic Irrigation and Debridement; Procedure: Open Arthrotomy with irrigation and debridement

INTERVENTIONS:
Procedure: Arthroscopic Irrigation and Debridement — Patients with confirmed septic arthritis treated with multiple small incisions to perform irrigation and debridement with partial synovectomy.
Procedure: Open Arthrotomy with irrigation and debridement — Patients with confirmed septic arthritis treated with a single large incision, open arthrotomy to perform irrigation and debridement with partial synovectomy.

SUMMARY:
Surgical excisional debridement is the mainstay of management in septic arthritis with necessary decompression, lavage, debridement, and partial synovectomy. However, there has been considerable debate over the optimal modality. Most surgeons perform an open arthrotomy or arthroscopic debridement, although serial aspiration can be considered as an option in very limited circumstances with patients who cannot tolerate surgery. While open arthrotomy has been often utilized, there has been an increasing number of proponents for arthroscopic treatment citing lower re-infection rates and better functional outcomes. However, there has been a lack of well-designed prospective studies comparing surgical treatment modalities for native knee septic arthritis. The goals of this present study are to determine if arthroscopic management of septic arthritis in the native knee resulted in a lower number of surgeries and a shorter length of stay compared to open arthrotomy. Secondary outcomes included differences in postoperative pain and improvements in Lysholm knee scores.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years old)
* Have a diagnosis of septic arthritis of the native knee (synovial WBC >50k or acrystalline elevated synovial WBC >25,000 with high clinical suspicion)
* Willingness to participate in the study

Exclusion Criteria:

* Unwilling to participate in the study
* Acrystalline elevated synovial WBC < 25,000
* Crystalline arthropathy with elevated synovial WBC but < 50,000
* Have a history of a prior knee prosthesis (hemiarthroplasty, total knee arthroplasty)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Number of surgeries to obtain lasting clinical resolution | Through time period of initial admission (days; expected under 14 days)
  The total number of surgeries performed during initial admission in order to obtain appropriate clinical response and resultant discharge on outpatient antibiotics.
Hospital length of stay | Through time period of initial admission (days; expected under 14 days)
  The total number of days in which the patient is initially admitted in order to obtain appropriate clinical response and resultant discharge on outpatient antibiotics.

SECONDARY OUTCOMES:
Post Operative Pain Scores | Through time period of initial admission (days; expected under 14 days)
  Daily morning and afternoon visual analogue scale reported by nursing staff. This value is reported on a scale of 0-10; a score of 0 indicates no pain while 10 indicates unbearable pain
Post Operative Opioid Use | Through time period of initial admission (days; expected under 14 days)
  All patients will have post operative pain medications which are to be utilized in a step wise manner for treating their pain. For example, if they are in minimal pain they will be given tylenol whereas unbearable pain will be treated with opioid analgesics. The average total post-operative opioid usage during initial admission will be reported as total morphine milligram equivalent.
Lysholm Knee Scale | Through anticipated follow up period of 3 month post operative appointment.
  The Lysholm score is a 100-point scoring system for examining a patient's knee-specific symptoms including mechanical locking, instability, pain, swelling, stair climbing, and squatting. The scoring is between 0-100 points. A score of <65 indicates poor knee function, 65-83 indicates fair knee function, 84-94 indicates a fair outcome, and 95-100 indicates excellent knee function. This scoring system will be obtained at 2 week, 6 week, and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Adler, MD, Study Director — Texas Tech University Health Sciences Center of El Paso
Locations (1):
- University Medical Center of El Paso, El Paso, Texas, United States

REFERENCES:
- [Background] Hunter JG, Gross JM, Dahl JD, Amsdell SL, Gorczyca JT. Risk factors for failure of a single surgical debridement in adults with acute septic arthritis. J Bone Joint Surg Am. 2015 Apr 1;97(7):558-64. doi: 10.2106/JBJS.N.00593. PMID 25834080
- [Background] Bohler C, Dragana M, Puchner S, Windhager R, Holinka J. Treatment of septic arthritis of the knee: a comparison between arthroscopy and arthrotomy. Knee Surg Sports Traumatol Arthrosc. 2016 Oct;24(10):3147-3154. doi: 10.1007/s00167-015-3659-8. Epub 2015 May 28. PMID 26017744
- [Background] Wirtz DC, Marth M, Miltner O, Schneider U, Zilkens KW. Septic arthritis of the knee in adults: treatment by arthroscopy or arthrotomy. Int Orthop. 2001;25(4):239-41. doi: 10.1007/s002640100226. PMID 11561499
- [Background] Aim F, Delambre J, Bauer T, Hardy P. Efficacy of arthroscopic treatment for resolving infection in septic arthritis of native joints. Orthop Traumatol Surg Res. 2015 Feb;101(1):61-4. doi: 10.1016/j.otsr.2014.11.010. Epub 2015 Jan 23. PMID 25623272

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT04786379/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT04786379/ICF_001.pdf